CLINICAL TRIAL: NCT02030990
Title: The Use of Intraoperative Mitomycin-C During Photorefractive Keratectomy and Its Effect on Postoperative Topical Steroid Requirements
Brief Title: The Use of MMC During PRK and Its Effect on Postoperative Topical Steroid Requirements
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Cason, MD., CDR US Navy, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NMCSD.2014.0032
Record Dates: First submitted 2013-12-20; First posted 2014-01-09 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Corneal Opacity
Keywords: photorefractive keratectomy; corneal haze; mitomycin-C; postoperative steroids
MeSH Terms: conditions — Corneal Opacity | interventions — Mitomycin; Fluorometholone

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mitomycin-C; 3 week FML steroid taper (Experimental): Mitomycin-C 0.01% will be administered intraoperatively during PRK for 15 seconds. The patient will take a 3 week fluorometholone 1% topical steroid taper.
  Interventions: Drug: Mitomycin-C; Drug: Fluorometholone 1% topical ocular steroid
- Mitomycin-C; 1 week FML steroid taper (Experimental): Mitomycin-C 0.01% will be administered intraoperatively during PRK for 15 seconds. The patient will take a 1 week of fluorometholone 1% topical steroid.
  Interventions: Drug: Mitomycin-C; Drug: Fluorometholone 1% topical ocular steroid
- No mitomycin-C; 8 week FML steroid taper (Active Comparator): No mitomycin-C will be administered during the procedure. Instead a sham application of salt solution will be given for 15 seconds. The patient will take 8 weeks of topical fluorometholone 1% topical steroid drop taper.
  Interventions: Drug: Fluorometholone 1% topical ocular steroid

INTERVENTIONS:
Drug: Mitomycin-C — 0.01% applied to cornea with a sponge during PRK
  Other Names: MMC
  Arms: Mitomycin-C; 1 week FML steroid taper; Mitomycin-C; 3 week FML steroid taper
Drug: Fluorometholone 1% topical ocular steroid — topical steroid drops applied to the cornea after PRK
  Other Names: FML

SUMMARY:
1. Purpose To evaluate the use of mitomycin-C (MMC) as an intraoperative adjunct during photorefractive keratectomy (PRK), its effect on postoperative healing and its ability to reduce the postoperative topical steroid course after the surgery.
2. Research Design This is a single-center, prospective, comparative cohort study.
3. Hypothesis There will not be a significant difference in the refractive corrections amongst the treatment groups, 12 months after surgery.
4. Objectives The primary study objective is to compare the effect of intraoperative MMC and a postoperative short topical steroid taper of 3 weeks, intraoperative MMC and a rapid topical steroid taper of 1 week, and a more commonly accepted postoperative regimen of a 2 month long topical steroid taper without any intraoperative MMC. The primary endpoint evaluated will be objective estimates of refractive error (WaveScan WaveFront™ System) at 12 months post-surgery. Secondarily, the extent of haze formation will be evaluated objectively using densitometry maps generated by automated Scheimpflug imaging of the cornea (Pentacam®). Furthermore, the subjective vision from the patients' perspective will be evaluated by questionnaires.

DETAILED DESCRIPTION:
1. Purpose To evaluate the use of mitomycin-C (MMC) as an intraoperative adjunct during photorefractive keratectomy (PRK), its effect on postoperative healing and its ability to reduce the postoperative topical steroid course after the surgery.
2. Research Design This is a single-center, prospective, comparative cohort study.
3. Hypothesis There will not be a significant difference in the refractive corrections amongst the treatment groups, 12 months after surgery.
4. Objectives The primary study objective is to compare the effect of intraoperative MMC and a postoperative short topical steroid taper of 3 weeks, intraoperative MMC and a rapid topical steroid taper of 1 week, and a more commonly accepted postoperative regimen of a 2 month long topical steroid taper without any intraoperative MMC. The primary endpoint evaluated will be objective estimates of refractive error (WaveScan WaveFront™ System) at 12 months post-surgery. Secondarily, the extent of haze formation will be evaluated objectively using densitometry maps generated by automated Scheimpflug imaging of the cornea (Pentacam®). Furthermore, the subjective vision from the patients' perspective will be evaluated by questionnaire.
5. Methodology At the Navy Refractive Surgery Center San Diego (NRSC SD), a total of 300 patients will be enrolled and randomly assigned to three cohorts. PRK will be performed in a standard fashion for all treatment groups. In the first two groups, intraoperative MMC 0.01% for a contact time of 15 seconds will be utilized. During the postoperative period, the first cohort will use the short steroid taper and the second cohort will use the rapid steroid taper. The third cohort will not receive any intraoperative MMC and will self-administer postoperative steroids, tapering for two months. All cohorts will be followed at 1 week, 1 month, 3 months, 6 months and 12 months after the procedure. Standard clinical measures of visual performance will be recorded. Since visually significant corneal haze is relatively rare, corneal densitometry will be used as an objective measure to detect subclinical corneal haze in addition to our usual subjective haze evaluation done by the clinical optometrists.

The patients will complete a voluntary questionnaire that evaluates their subjective impression of the refractive surgery, their recovery and their outcomes. Specifically, the patient will report the use of refractive correction, usefulness of the surgery at work, dry eye complaints, and subjective appraisal of their vision.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty male or female, of any race, and at least 21 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 is intended to ensure documentation of refractive stability.
2. Manifest spherical equivalent (MSE) from +3.00 D to -11.0D with refractive cylinder of up to 3.00 D.
3. Best spectacle corrected visual acuity of 20/25 or better in both eyes.
4. Stable spectacle refraction, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50 D during the six-month period immediately preceding the baseline examination for myopic patients and 0.75 for hyperopic patients.
5. Contact lens use: Soft contact lenses must have been removed at least two (2) weeks prior to baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least four (4) weeks prior to baseline measurements.
6. Strong motivation for attending the follow-up visits and orders to remain in the area for the duration of at least twelve months of follow up.
7. Consent of the subject's command to participate in the study.
8. Access to transportation to meet follow up requirements.

Exclusion Criteria:

1. Aviators.
2. Female subjects who are pregnant, breast-feeding, or intend to become pregnant during the course of the study.
3. Concurrent topical or systemic medications which may impair healing, including corticosteroids, antimetabolites, isotretinoin, (Accutane™), amiodarone hydrochloride (Cordarone™), and/or sumatriptan (Imitrex™).
4. Medical conditions which, in the judgment of the investigator, may impair healing, including but not limited to thyroid disorders and diabetes.
5. Active ophthalmic disease, neovascularization of the cornea within 1 mm of the intended ablation zone, or lens opacity.
6. Evidence of glaucoma or an intraocular pressure greater than 22 mm Hg at baseline.
7. Evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
8. Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
9. Any physical or mental impairment which would preclude participation in any of the examinations, such as inability to give verbal responses to eye charts.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Refractive Error | 12 months
  Objective refractive error with Wavescan Aberrometry

SECONDARY OUTCOMES:
Refractive Error | 12 months
  Manifest refraction by patient subjective report
Corneal haze | 12 months
  Subjective grading by slit lamp examiner
Corneal haze | 12 months
  Subclinical objective measurement of corneal haze by Pentacam densitometry

CONTACTS AND LOCATIONS:
Overall Officials: John B Cason, M.D., Principal Investigator — United States Naval Medical Center, San Diego; Donna Murdoch, Ph.D., Study Director — Navy Warfighter Refractive Surgery San Diego
Locations (1):
- Navy Warfighter Refractive Surgery Center, San Diego, California, United States